CLINICAL TRIAL: NCT04799379
Title: Evaluation of Microporous Polysaccharide Hemospheres (MPH) Agent in Preventing Postoperative Complications After Rectal Surgery (EPHAS Study).
Brief Title: Microporous Polysaccharide Hemospheres (MPH) Improving Outcome After Rectal Surgery
Acronym: EPHAS
Status: Completed | Type: Observational
Sponsor: Grupo Español de Rehabilitación Multimodal (Other)
Collaborators: Universidad de Zaragoza (Other); Aragon Health Science Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: GERM-EPHAS
Record Dates: First submitted 2021-02-26; First posted 2021-03-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Sepsis
Keywords: Rectal surgery; Pelvic drain; microporous polysaccharide hemospheres
MeSH Terms: interventions — 5,10-dihydro-5-methylphenazine; Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: microporous polysaccharide hemospheres (MPH) agent in rectal surgery — Use of microporous polysaccharide hemospheres (MPH) agent in patients after rectal surgery to avoid pelvic collections and the use of any drain

SUMMARY:
Multi-center, prospective, cohort study, of patients scheduled for elective rectal surgery who received absorbable hemostatic powder to assess whether it can improve patient postoperative outcomes, reduce usage of drains and prove to be cost-effective. This cohort will be compared to a previously studied cohort using drains (Power and IMPRICA study) with comparable patient characteristics.

The primary endpoint of the study is: postoperative pelvic sepsis within 60 postoperative days including anastomotic leakage, pelvic abscess and peritonitis.

Secondary endpoints: postoperative morbidities, rate of reoperation and length of hospitalization.

DETAILED DESCRIPTION:
Multimodal surgical rehabilitation, also known as Enhanced Recovery After Surgery, entails the application of a series of perioperative procedure measures and strategies aimed at patients who are going to undergo a surgical procedure with the objective of reducing secondary stress caused by the surgical intervention and thus achieve enhanced recovery of the patient and decrease complications and mortality.

ERAS protocols are care programs based on scientific evidence, encompassing all aspects of patient care and requiring multidisciplinary management, with the participation of diverse specialists1. Starting at the diagnosis, their aim is to recognize patients' individual needs to optimize their treatment before, during and after surgery. The close collaboration of all specialists participating in the process, as well as of the actual patients and their relatives has proved to be essential.

The Multimodal Rehabilitation Programmes (MRP) or Enhanced Recovery Programmes (ERAS) review traditional perioperative procedure practices, evaluating the specific key points of each type of surgery and analysing their scientific evidence. MRPs have shown, in cents that have routinely adopted them, a significant improvement in the patient's quality of life. Furthermore, MRPs significantly reducing the hospital stay and potential complications associated with hospitalisation2, being the anastomotic leak (AL) the most serious of them.

Total mesorectal excision (TME) and bowel restoration is currently the standard treatment for middle to low rectal cancer. However, TME has been shown to be associated with high anastomotic leakage with a reported incidence of up to 24%, reaching 50% when clinically silent radiographic leaks are considered3.

Despite a large number of studies in the literature that have investigated risk factors, the fundamental causes of AL remain unclear. In this sense, according to enhanced recovery after surgery (ERAS) protocols4, pelvic drain should not be used routinely as it may cause patient discomfort and prolong hospitalization. Moreover, drain itself is also a potential site of infection especially if open or passive drainage system is used.

Even based in the best available evidence, ERAS protocols have important implementation problems because they have to put up with traditional attitudes. In this sense, many surgeons still advocate the use of a prophylactic pelvic drain because they believe that fluid collection in the pelvis could be a potential source of contamination and thereby weakening anastomotic integrity and healing.

In a recent study from the Spanish group GERM2, avoidance of drains was achieved only in 34.7% of patients undergoing elective colorectal surgery. ERAS centres had a greater avoidance of drains vs non-ERAS centres (38.6% vs 28.3%), although most patients still received drains. More relevant, avoidance of drainage was associated with a significant reduction in moderate to severe complications.

We believe that it is more than justified to try new options that help surgeons reduce the use of drains. One of these, is the use of hemostatic agents. Some topical hemostats may theoretically be of benefit due to its claimed lymphostatic properties.

Published data for this is sparse, but some studies, have shown statistically significant reduction of fluid collection after using Arista®AH5.

Arista is a plant-based, flowable powder engineered to rapidly dehydrate blood, enhancing clotting on contact. Arista facilitates the formation of a highly resilient, natural clot within just a few minutes regardless of the patient's coagulation status. Arista® is fully absorbable within 24 to 48 hours of application, and because Arista degrades rapidly, it does not promote infection.

This study has been designed to support the working hypothesis that Arista® placed intraoperatively into the dissected pelvic area could reduce sepsis and postoperative anastomotic leakage. We choose to study Arista® for a theoretical reason: it contains microporous polysaccharide hemospheres (MPHs). MPHs not only activate the coagulation cascade but they cause tissue desiccation which presumably seals capillaries and could theoretically also seal small lymph vessels left open by electrosurgical devices.

Study assumptions: Arista spread on the pelvic floor at the end of surgery may allow to

1. close small holes and prevent fluid from penetrating into the pelvic floor, thereby avoiding AL
2. facilitate the avoidance of drains

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (aged >18 years) with a diagnosis of malignant rectal cancer who are scheduled for radical surgery (anterior resection). Informed consent will be obtained from all subjects, who will participate in the study voluntarily.

Exclusion Criteria:

* Patient refusal, patients undergoing emergency surgery, patients under 18 years of age, existence of other concomitant surgical processes. Previous chemo-radiotherapy. Ileostomy or colostomy. Patients that have receive a drain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged >18 years) with a diagnosis of malignant rectal cancer who are scheduled for radical surgery. This study will be conducted in 12 Spanish general hospitals, which are selected on the basis of having established an enhanced recovery protocol that complies with the recommendations of the Aragon Health Sciences Institute (IACS) and Spanish National Health Service (https://portal.guiasalud.es/wpcontent/uploads/2019/10/viaclinica-rica_english.pdf)
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
postoperative pelvic sepsis including anastomotic leakage, pelvic abscess and peritonitis. | 60 days
  % patients with organ-space infection or anastomotic leak

SECONDARY OUTCOMES:
postoperative morbidities | 60 days
  % Patients with at least one complication related to the surgical intervention
rate of reoperation | 60 days
  % patients requiring reoperation for any cause
Hospital stay | 60 days
  Total number of days of stay included pre and postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Blanco, PhD, Principal Investigator — Hospital de la Ribera
Locations (5):
- Spain (5):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital de la RIBERA, Alzira, Valencia
  - Hospital Jimenz diaz, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ruiz-Tovar J, Sanchez-Santos R, Martin-Garcia-Almenta E, Garcia Villabona E, Hernandez AM, Hernandez-Matias A, Ramirez JM; grupo de Trabajo de Cirugia Bariatrica del Grupo Espanol de Rehabilitacion Multimodal (GERM). Enhanced recovery after bariatric surgery. Cir Esp (Engl Ed). 2019 Dec;97(10):551-559. doi: 10.1016/j.ciresp.2019.05.003. Epub 2019 Jun 18. English, Spanish. PMID 31221424
- [Background] Ripolles-Melchor J, Ramirez-Rodriguez JM, Casans-Frances R, Aldecoa C, Abad-Motos A, Logrono-Egea M, Garcia-Erce JA, Camps-Cervantes A, Ferrando-Ortola C, Suarez de la Rica A, Cuellar-Martinez A, Marmana-Mezquita S, Abad-Gurumeta A, Calvo-Vecino JM; POWER Study Investigators Group for the Spanish Perioperative Audit and Research Network (REDGERM). Association Between Use of Enhanced Recovery After Surgery Protocol and Postoperative Complications in Colorectal Surgery: The Postoperative Outcomes Within Enhanced Recovery After Surgery Protocol (POWER) Study. JAMA Surg. 2019 Aug 1;154(8):725-736. doi: 10.1001/jamasurg.2019.0995. PMID 31066889
- [Background] Cavaliere D, Popivanov G, Cassini D, Cirocchi R, Henry BM, Vettoretto N, Ercolani G, Solaini L, Gerardi C, Tabakov M, Tomaszewski KA. Is a drain necessary after anterior resection of the rectum? A systematic review and meta-analysis. Int J Colorectal Dis. 2019 Jun;34(6):973-981. doi: 10.1007/s00384-019-03276-4. Epub 2019 Apr 25. PMID 31025093
- [Background] Luong J, Milanese E, Fortino J, Vetto JT. Reduction of lymphocele rate in patients undergoing sentinel node biopsy for melanoma by intraoperative placement of plant-based hemostatic powder: Results of a prospective trial. Am J Surg. 2019 May;217(5):878-881. doi: 10.1016/j.amjsurg.2019.02.016. Epub 2019 Feb 14. PMID 30799018
- [Background] Grupo de trabajo. Vía Clínica de Recuperación Intensificada en Cirugía Abdominal (RICA). Vía clínica de recuperación intensificada en cirugía abdominal (RICA) Ministerio de Sanidad, Servicios Sociales e Igualdad. Instituto Aragonés de Ciencias de la Salud. 2014 Available from: http://portal.guiasalud.es/contenidos/iframes/documentos/ opbe/2015-07/ViaClinica-RICA.pdf